CLINICAL TRIAL: NCT02475902
Title: Health in Motion- Interactive Exercises for Safer Mobility
Acronym: HiM-O
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blue Marble Rehab Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TC053013
Record Dates: First submitted 2015-06-15; First posted 2015-06-19 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Accidental Falls
Keywords: prevention and control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer guided home exercise program (Experimental): A laptop computer & MS Kinect camera will be connected to a 40" TV to deliver guided fall prevention exercises. Research staff will train the participants in the use of the computerized program and be supervised performing the exercises during the instruction period. Then participants will be instructed to exercise 3 times per week for 4 weeks. Half of the participants will begin the study with the computerized version of the home exercise program while the other half begins with the paper booklet version of the home exercise program. After one month the arms will cross over.
  Interventions: Behavioral: Computer guided home exercise program
- Paper guided home exercise program (Active Comparator): A paper booklet with pictures and written instructions, and an exercise log for the home exercise program will be given to half of the participants. Participants will be carefully instructed in performing the exercises correctly and then asked to perform the exercises 3 times per week for one month. Participants who began the study with the paper exercise program will switch to the computerized version of the exercise program for the second month.
  Interventions: Behavioral: Paper guided home exercise program

INTERVENTIONS:
Behavioral: Computer guided home exercise program — Participants will follow a computerized fall prevention home exercise program with MS Kinect camera tracking 3 times per week for one month.
  Arms: Computer guided home exercise program
Behavioral: Paper guided home exercise program — Participants will follow a fall prevention home exercise program outlined in a paper booklet 3 times per week for one month.
  Arms: Paper guided home exercise program

SUMMARY:
The participants will complete a series of balance assessments with a licensed physical (PT) or occupational therapist (OT) or qualified research assistant (RA) at Blue Marble Game Co or in their respective homes at the start of the study, at crossover and upon completion of the study. During this study a PT, OT, or RA trained in fall risk management will supervise the instruction and practice by participants of the home exercise programs during the initial 2-3 hour introduction to the study activities. Participants will be asked to exercise 3/week for one month then crossover to the alternative exercise program and exercise 3/week for a second month.

DETAILED DESCRIPTION:
The participants will complete a series of balance assessments with a licensed physical (PT) or occupational therapist (OT) or qualified research assistant (RA) at Blue Marble Game Co or in their respective homes at the start of the study, at cross over and upon completion of the study. During this study a PT, OT, or RA trained in fall risk management will supervise the instruction and practice by participants of the home exercise programs during the initial 2-3 hour introduction to the study activities. Participants will be asked to exercise 3/week for one month then crossover to the alternative exercise program and exercise 3/week for a second month. The PT, OT, or RA will determine that the participant is competent to perform the home exercise programs safely, with no more than a normal risk of falls or withdraw the participant from the study. The participant's score on the standard version of the Falls Risk Questionnaire, Single Leg Stance Test, and Chair Rise Test will be recorded and stored on a password protected computer in a locked office. Once the data has been stored electronically, paper data collection sheets will be placed in a confidential bin for shredding. Exercise Data will be captured using a) the Health In Motion software via the Kinect Sensor and stored on the Blue Marble secure server and b) via a daily exercise log provided to the participant in paper form.

ELIGIBILITY:
Inclusion Criteria:

* Health status: Individuals medically stable and have no medical condition that would affect their participation in group discussion or that would affect their ability to perform the balance assessments or balance exercises. The participants for Study 1 and 2 are required to walk 500 feet independently without an assistive device (e.g. walker, cane or person).
* Gender: 50%/50% male and female
* Ability to speak/read English fluently (focus group will be conducted in English & art work will have English text)
* For Study 1 and 2, the participant must have had less than 2 falls in the past 12 months.

Exclusion Criteria:

* History of seizure activity when watching TV or when playing video games.
* Unable to learn to use the technology safely without direct supervision.
* Insufficient clear, safe exercise space in the home with internet access.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change in Timed up and go test score | baseline, 1 month, 2 months

SECONDARY OUTCOMES:
Fear of Falling Avoidance Behavior Questionnaire | baseline, 1 month, 2 months
Functional Reach Test | baseline, 1 month, 2 months
Berg Balance Scale | baseline, 1 month, 2 months
Health Related Quality of Life: SF-36 | baseline, 1 month, 2 months

OTHER OUTCOMES:
System Usability Scale (Questionnaire) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Flynn, PhD, Principal Investigator — Blue Marble Rehabilitation, Inc.